CLINICAL TRIAL: NCT05993429
Title: Diagnostic Efficacy of Endoscopic Ultrasound-guided Fine-needle Aspiration/Biopsy Versus Endoscopic Retrograde Cholangiopancreatography With or Without Peroral Cholangioscopy Targeted Biopsy for Suspected Hilar Cholangiocarcinoma: an Open Multicenter Prospective Study
Brief Title: Diagnostic Efficacy of EUS-FNA/B Versus ERCP With or Without POCS-TB in Patients With Suspected Hilar Cholangiocarcinoma
Status: Completed | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); First Affiliated Hospital of Guangxi Medical University (Other); LanZhou University (Other); Beijing Friendship Hospital (Other); Binzhou Medical University (Other); Shandong Provincial Hospital (Other Government); Shandong Province Third hospital (Other); Sir Run Run Shaw Hospital (Other); The Third Xiangya Hospital of Central South University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 2023SDU-QILU-3
Record Dates: First submitted 2023-07-13; First posted 2023-08-15 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2024-08

CONDITIONS: Klatskin Tumor; Cholangiocarcinoma; Biopsy, Fine-Needle; Endoscopic Retrograde Cholangiopancreatography
MeSH Terms: conditions — Klatskin Tumor; Cholangiocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EUS-FNA/B group; ERCP with or without POCS-TB group: EUS-FNA/B group: Patients with suspected hilar cholangiocarcinoma who were considered suitable for obtaining histopathological diagnosis by EUS-FNA/B by experts
  Interventions: Diagnostic Test: The sampling method selected in patients with suspected hilar cholangiocarcinoma
- ERCP with or without POCS-TB group: ERCP with or without POCS-TB group: Patients with suspected hilar cholangiocarcinoma who were considered suitable for obtaining histopathological diagnosis by ERCP with or without POCS-TB by experts
  Interventions: Diagnostic Test: The sampling method selected in patients with suspected hilar cholangiocarcinoma

INTERVENTIONS:
Diagnostic Test: The sampling method selected in patients with suspected hilar cholangiocarcinoma — The appropriate sampling approach was selected as EUS-FNA/B or ERCP with or without POCS-TB based on experts' overall evaluation. This study will compare the histopathological diagnosis of the selected sampling method with the final diagnosis.

SUMMARY:
This is an observational study with a prospective cohort design. This study enrolled patients with suspected hilar cholangiocarcinoma on imaging. This study aims to evaluate the histopathological diagnostic efficacy of endoscopic ultrasound-guided fine-needle aspiration/biopsy (EUS-FNA/B) and endoscopic retrograde cholangiopancreatography (ERCP) with or without peroral cholangioscopy targeted biopsy (POCS-TB) in patients with suspected hilar cholangiocarcinoma. In addition, the incidence of complications was compared between the EUS-FNA/B and ERCP with or without POCS-TB. The impact of the histopathological diagnosis on survival outcomes in patients with suspected hilar cholangiocarcinoma was evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old;
2. Newly diagnosed patients with suspected hilar cholangiocarcinoma on imaging examination

Exclusion Criteria:

1. Patients with a definite diagnosis of cholangiocarcinoma by imaging (enhanced CT, MRI, or MRCP) and surgical candidacy within 3 months;
2. Patients scheduled for liver transplantation;
3. Patients with previous gastroduodenal diversion or biliary surgery;
4. Patients with hilar bile duct stenosis caused by tumor or lesion outside the bile duct;
5. Pregnant or lactating women;
6. Patients who cannot tolerate intravenous general anesthesia due to various reasons;
7. Patients with severe coagulation dysfunction, or patients who cannot stop antiplatelet/anticoagulant therapy for a short time and are unsuitable for low molecular weight heparin replacement therapy;
8. Patients who refused to sign informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with suspected hilar cholangiocarcinoma who were considered suitable for obtaining histopathological diagnosis by EUS-FNA/B or ERCP with or without POCS-TB by experts
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-08-14 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
The diagnostic value of EUS-FNA/B versus ERCP with or without POCS-TB in diagnosing hilar cholangiocarcinoma | 2023-08-14 to 2027-08-01
  The diagnostic value was assessed by sensitivity, specificity, accuracy, and positive and negative predictive values.

SECONDARY OUTCOMES:
The incidence of complications | 2023-08-14 to 2027-08-01
  The incidence of complications after EUS-FNA/B versus ERCP with or without POCS-TB
The cost-effectiveness ratio | 2023-08-14 to 2027-08-01
  The cost-effectiveness ratio of EUS-FNA/B versus ERCP with or without POCS-TB in the diagnosis of hilar cholangiocarcinoma
The emergency readmission time | 2023-08-14 to 2027-08-01
  The emergency readmission time of EUS-FNA versus ERCP with or without POCS-TB
The proportion of tissue deemed adequate for cytological or histological analysis obtained by EUS-FNA/B and ERCP with or without POCS-TB. | 2023-08-14 to 2027-08-01
  The proportion of tissue deemed adequate for cytological or histological analysis obtained by EUS-FNA/B and ERCP with or without POCS-TB.
The number of participants whose visual diagnosis by the new generation of Eye Max cholangioscopy was consistent with the pathological and final diagnoses, respectively. | 2023-08-14 to 2027-08-01
  The number of participants whose visual diagnosis by the new generation of Eye Max cholangioscopy was consistent with the pathological and final diagnoses, respectively.
The number of participants whose management was affected by the new generation of Eye Max cholangioscopy visual diagnosis. | 2023-08-14 to 2027-08-01
  The number of participants whose management was affected by the new generation of Eye Max cholangioscopy visual diagnosis.
The incidence rate of needle tract metastasis by EUS-FNA/B | 2023-08-14 to 2027-08-01
  The incidence rate of needle tract metastasis by EUS-FNA/B
The number of participants whose further treatment strategies were impacted by preoperative pathological diagnosis. | 2023-08-14 to 2027-08-01
  The number of participants whose further treatment strategies were impacted by preoperative pathological diagnosis.
The number of participants whose survival outcomes were impacted by preoperative pathological diagnosis. | 2023-08-14 to 2027-08-01
  The number of participants whose survival outcomes were impacted by preoperative pathological diagnosis.
Maximum lesion size | 2023-08-14 to 2027-08-01
  Maximum lesion size on EUS
Lesion shape | 2023-08-14 to 2027-08-01
  Lesion shape (ovoid-to-round, irregular) on EUS.
Lesion composition | 2023-08-14 to 2027-08-01
  Lesion composition (cystic, partially cystic, solid) on EUS.
Lesion margin | 2023-08-14 to 2027-08-01
  Lesion margin (ill-defined, microlobulated/spiculated, well-defined) on EUS.
Lesion echogenicity | 2023-08-14 to 2027-08-01
  Lesion echogenicity (hyperechoic intensity, isoechoic intensity, hypoechoic intensity) on EUS.
Lesion heterogeneity | 2023-08-14 to 2027-08-01
  Lesion heterogeneity on EUS.
Lesion growth pattern | 2023-08-14 to 2027-08-01
  Lesion growth pattern on EUS.
Lesion blood flow | 2023-08-14 to 2027-08-01
  Lesion blood flow (none, poor, moderate, rich) on EUS.
Lesion elastography | 2023-08-14 to 2027-08-01
  Lesion elastography (stiff, moderate, soft, unvalued) on EUS.

CONTACTS AND LOCATIONS:
Overall Officials: Ning Zhong, MD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No